CLINICAL TRIAL: NCT03200925
Title: The Effect of Video Education on Skin-to-Skin at the Time of Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kettering Health Network (Other)
Collaborators: Ohio University (Other)
Responsible Party: Principal Investigator, Catherine Caponero, Principal Investigator, Kettering Health Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1078384-2
Record Dates: First submitted 2017-06-25; First posted 2017-06-27 (Actual); Results first posted 2019-07-22 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Kangaroo Care; Video; Prenatal Education; Skin-to-skin
Keywords: video; skin-to-skin; kangaroo care; prenatal education

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will not know which arm of the trial they will be apart of until after they have consented to participate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - no video group (No Intervention): Group A will be asked a short survey:
  * their intention to practice skin to skin at the time of delivery
  * if they participated in skin to skin in a previous pregnancy
  * if they had any formal education about skin to skin
  * if they did have formal education was it either
    * a.) Provided at a prenatal appointment,
    * b.) A formal class led by either a nurse or a lactation consultant.
  We will also look at patient's medical record number, age, gestational age, any pregnancy complications, race, type of insurance, and the number of times the patient has been pregnant. We will also examine data that is already collected by this hospital after delivery regarding skin to skin. This includes gestational age in weeks at the time of delivery, 5 minute APGAR, delivery date/time, skin to skin initiation time, skin to skin end time, delivery to skin to skin duration (minutes), and skin to skin duration (minutes).
- Group B - video group (Experimental): Group B will be asked the same short survey as group A.
  The patient would then immediately watch "Jumping into Kangaroo Care", and then immediately take the post survey which would ask if they intended to practice skin to skin at the time of delivery.
  We will also look at patient's medical record number, age, gestational age, any pregnancy complications, race, type of insurance, and the number of times the patient has been pregnant. We will also examine data that is already collected by this hospital after delivery regarding skin to skin. This includes gestational age in weeks at the time of delivery, 5 minute APGAR, delivery date/time, skin to skin initiation time, skin to skin end time, delivery to skin to skin duration (minutes), and skin to skin duration (minutes).
  Interventions: Other: "Jumping into Kangaroo Care" - a video created by the Ohio Department of Health

INTERVENTIONS:
Other: "Jumping into Kangaroo Care" - a video created by the Ohio Department of Health — The video is 8 minutes and 52 seconds in length. The video discusses the benefits and logistics of Kangaroo Care from professional's perspectives and from new mother's perspectives.
  Arms: Group B - video group

SUMMARY:
The main purpose of this study is to determine the effect of prenatal video education on pregnant women's intention to practice and actual practice of skin to skin contact (SSC) after birth. This study hypothesizes that education in video format will increase patients knowledge about skin to skin in a way that will make them consider participating in skin to skin immediately after birth.

Therefore the end point for this study is intention to participate in SCC measured by a single questionnaire item "Do you plan on participating in skin to skin (or kangaroo care) immediately after birth?" Our secondary end-point will measure whether or not the patient was able to participate in skin to skin within five minutes of delivery.

All study participants will complete a short survey about their intention of practicing skin to skin after birth upon admission for delivery. Half of the study participants will only complete the brief survey. The other half of study participants will then watch a short video about skin to skin and complete one follow up question regarding their intention to practice skin to skin at the time of delivery. All patients will be followed until after delivery to determine if they were able to participate in skin to skin after delivery.

DETAILED DESCRIPTION:
Despite strong support of breastfeeding by organizations such as the American Academy of Pediatrics, the American Congress of Obstetricians and Gynecologists, and the American Academy of Family Physicians, the rate of breastfeeding initiation at the time of delivery and continuation at 6 months postpartum is below the Center of Disease Prevention's Healthy People 2010 goals (1). UNICEF and the World Health Organization (WHO) have estimated that if all babies were breastfed for a minimum of the first six months of their lives, the rate of morbidity and malnutrition would significantly decrease all over the world (2). The benefits of breastfeeding are numerous for both mothers and infants, with infants obtaining optimal nutrition and passive immunity, and mothers obtaining a more rapid return of postpartum uterine tone, postpartum weight loss, delay of ovulation, and decreased risk of breast, ovarian, and endometrial cancers (3). As a result of this information, in 1991 WHO and UNICEF launched the Baby-Friendly Hospital Initiative (BFHI) to encourage proper infant feeding practices starting at birth. It is based on ten steps, which the hospital must meet and maintain to obtain certification. In support of Step Four of the BFHI to "help mothers initiate breastfeeding within one hour of birth," the skin-to-skin variation of Kangaroo Mother Care was initiated (4).

Kangaroo position, or skin to skin contact (SSC) on a mother's chest, provides thermoregulation, physiological stability, appropriate stimulation, and encourages bonding and breastfeeding (5). In fact, early SSC was significantly associated with type of feeding at discharge through 3 months postpartum (6). Regrettably, according to the American Academy of Pediatrics, some obstacles to SSC and breastfeeding include insufficient prenatal education, disruptive obstetrical practices, and a lack of family and societal support (7). Delivery room and postpartum hospital routines may also significantly disrupt early maternal-infant interactions (8). These barriers to breastfeeding and SSC are more prevalent amongst vulnerable groups, which includes low income, low educational level, and black populations. While effective initiatives such as BFHI are present in hospital settings, guidelines for primary care based interventions originating in a clinician's office currently do not exist (3). Through encouraging education regarding SSC before the time of delivery, patients can actively participate in SSC during delivery and advocate for early SSC (9).

Education can easily influence behavior habits and does not need to require special difficulties on behalf of providers (9). In fact, educational programs have the single greatest effect of any single intervention on both initiation and short term duration for breastfeeding (3). Women who attended breastfeeding classes with lactation consultants - with or without video supplementation - had significantly increased breastfeeding at six months when compared to controls (1). Currently, common office practices include provision of written materials and discharge packets. Neither practice has been shown to be effective in increasing rates of breastfeeding. On the contrary, discharge packets have been shown to reduce the rates of breastfeeding (3). Ideally, breastfeeding education would use both individual or group sessions where both benefits of breastfeeding and SSC would be discussed (10). However, in a busy clinic setting filled with a vulnerable patient population, having the ability to get to extra educational classes is not always an option.

Regardless of amount of prenatal education provided, Southview Medical Center will study participating patients at the time of admission for delivery who watch an 8 minutes 52 second patient education DVD titled "Jumping into Kangaroo Care" by the Ohio Department of Health. Of importance, studies so far have shown no clear pattern for the outcome of breastfeeding in respect to intervention timing (7). In an analysis regarding video modeling, patients who viewed videotapes regarding treatment options had a greater understanding of the risks and benefits of those choices and were more apt to be active participants in decision making (11). Audio-visual material can also be entertaining and can be used by those who have limited literacy. Moreover, the information provided to patients on video has the advantage of being repeatable and consistent, which would allow us to provide the same information to all of our patients (12). By educating patients in a video format at the beginning of their delivery admission, patients will have time to formulate questions and opinions to help them engage in an active dialogue with the staff that will be preforming the delivery. The goal of educating mothers is not only to increase their knowledge and skills but also to influence their attitudes (13). By providing a video which models SSC to all non-emergent anticipated vaginal deliveries upon admission to the hospital, the investigators' hope is to encourage patients to actively participate in SSC at the time of delivery and become their own advocates.

The main purpose of this study is to determine the effect of prenatal video education on pregnant women's intention to practice SSC after birth. This study is critical as quality measures for Southview Medical Center for quarter one of 2017 showed that the hospital has only been 50% successful at initiating skin to skin in vaginal deliveries after 37 weeks gestation with a 5 minute APGAR of 7. The hospital's goal per BFHI is 82%. The investigators' hypothesis is that 30% or more women who did not plan to use SCC would indicate their intention to use SSC post-intervention as compared to those who did not receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at Southview Medical Center
* Over the age of 18
* Anticipating a vaginal delivery within one week of admission to labor and delivery
* English speaking
* Greater than 37 weeks gestation

Exclusion Criteria:

* Not female
* Not pregnant
* Less than 37 weeks gestation
* A scheduled cesarean section
* Unstable medical status
* Expecting an unstable baby requiring medical resuscitation
* Under the age of 18
* Non-English speaking requiring translation services

If a patient has a baby with a 5 minute APGAR less than 7 at the time of delivery or needs to proceed to the operating room for cesarean delivery, the patient would not be included in data collection regarding skin to skin at the time of delivery. For this group, only intention would be measured

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Caponero, DO, Principal Investigator — Kettering Health Network
Locations (1):
- Southview Medical Center, Centerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen IM, Krueger MV, Carney LM, Graham JA. Prenatal breastfeeding education and breastfeeding outcomes. MCN Am J Matern Child Nurs. 2008 Sep-Oct;33(5):315-9. doi: 10.1097/01.NMC.0000334900.22215.ec. PMID 18758336
- [Background] Burgio MA, Lagana AS, Sicilia A, Prosperi Porta R, Porpora MG, Ban Frangez H, DI Venti G, Triolo O. Breastfeeding Education: Where Are We Going? A Systematic Review Article. Iran J Public Health. 2016 Aug;45(8):970-977. PMID 27928522
- [Background] Guise JM, Palda V, Westhoff C, Chan BK, Helfand M, Lieu TA; U.S. Preventive Services Task Force. The effectiveness of primary care-based interventions to promote breastfeeding: systematic evidence review and meta-analysis for the US Preventive Services Task Force. Ann Fam Med. 2003 Jul-Aug;1(2):70-8. doi: 10.1370/afm.56. PMID 15040435
- [Background] Baby-Friendly USA. "Guidelines and Evaluation Criteria for Facilities Seeking Baby-Friendly Designation." Albany, NY: Baby-Friendly USA. 2016
- [Background] Charpak N, Ruiz JG. Latin American Clinical Epidemiology Network Series - Paper 9: The Kangaroo Mother Care Method: from scientific evidence generated in Colombia to worldwide practice. J Clin Epidemiol. 2017 Jun;86:125-128. doi: 10.1016/j.jclinepi.2016.05.019. Epub 2016 Oct 17. PMID 27765653
- [Background] Vila-Candel R, Duke K, Soriano-Vidal FJ, Castro-Sanchez E. Affect of Early Skin-to-Skin Mother-Infant Contact in the Maintenance of Exclusive Breastfeeding: Experience in a Health Department in Spain. J Hum Lact. 2018 May;34(2):304-312. doi: 10.1177/0890334416676469. Epub 2017 Jan 18. PMID 28099044
- [Background] Chung M, Raman G, Trikalinos T, Lau J, Ip S. Interventions in primary care to promote breastfeeding: an evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2008 Oct 21;149(8):565-82. doi: 10.7326/0003-4819-149-8-200810210-00009. PMID 18936504
- [Background] Moore ER, Anderson GC, Bergman N. Early skin-to-skin contact for mothers and their healthy newborn infants. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003519. doi: 10.1002/14651858.CD003519.pub2. PMID 17636727
- [Background] Martinez-Galiano JM, Delgado-Rodriguez M. Influence of an education program of pregnant women on delivery. J Matern Fetal Neonatal Med. 2014 May;27(7):719-23. doi: 10.3109/14767058.2013.836486. Epub 2013 Sep 25. PMID 23962180
- [Background] Krouse HJ. Video modelling to educate patients. J Adv Nurs. 2001 Mar;33(6):748-57. doi: 10.1046/j.1365-2648.2001.01716.x. PMID 11298212
- [Background] Abu Abed M, Himmel W, Vormfelde S, Koschack J. Video-assisted patient education to modify behavior: a systematic review. Patient Educ Couns. 2014 Oct;97(1):16-22. doi: 10.1016/j.pec.2014.06.015. Epub 2014 Jul 5. PMID 25043785
- [Background] Shealy KR, Li R, Benton-Davis S, Grummer-Strawn LM. The CDC Guide to Breastfeeding Interventions. Atlanta: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, 2005
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B - Video Group: Group B will be asked the same short survey as group A. The patient would then immediately watch "Jumping into Kangaroo Care", and then immediately take the post survey which would ask if they intended to practice skin to skin at the time of delivery.We will also look at patient's medical record number, age, gestational age, any pregnancy complications, race, type of insurance, and the number of times the patient has been pregnant. We will also examine data that is already collected by this hospital after delivery regarding skin to skin. This includes gestational age in weeks at the time of delivery, 5 minute APGAR, delivery date/time, skin to skin initiation time, skin to skin end time, delivery to skin to skin duration (minutes), and skin to skin duration (minutes).
Period: Overall Study
Arm/Group | Group A - no Video Group | Group B - Video Group
Started | 120 | 120
Completed | 120 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - no Video Group | Group B - Video Group | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (5.5) | 27 (5.1) | 27 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 120 | 240
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 90 | 98 | 188
  African American | 22 | 12 | 34
  Hispanic | 4 | 1 | 5
  Other | 4 | 9 | 13
Primiparous [Count of Participants; unit: Participants] | 53 | 55 | 108
Private Insurance [Count of Participants; unit: Participants] | 55 | 58 | 113
Medicaid [Count of Participants; unit: Participants] | 61 | 58 | 119
Comorbidities [Count of Participants; unit: Participants]
  Chronic Hypertension | 5 | 3 | 8
  Gestational Hypertension | 6 | 10 | 16
  Preeclampsia | 3 | 2 | 5
  Gestational Diabetes Mellitus | 4 | 9 | 13
  Asthma | 10 | 10 | 20
  Neurologic Disease | 4 | 1 | 5
  Hematologic Disease | 13 | 9 | 22
  Other Medical Comorbitities | 40 | 42 | 82
Obstetric Measures [Count of Participants; unit: Participants]
  Spontaneous Vaginal Delivery | 84 | 89 | 173
  Vacuum Delivery | 11 | 9 | 20
  Low Transverse Cesarean Delivery | 25 | 22 | 47
Gestational Age (weeks) [Mean (Full Range); unit: weeks] | 39 [37 to 41] | 39 [37 to 41] | 39 [37 to 41]
5 Minute APGAR Score [Median (Full Range); unit: units on a scale] — APGAR is a standardized way to evaluate a baby's health and it stands for "Appearance, Pulse, Grimace, Activity, and Respiration." Each of the five categories are scored on a scale of 0 to 2, with 2 being the best score. The scores of the individual categories are then added together to create a total score which ranges from 0 to 10, with 10 being the best total score. The APGAR scoring system is typically utilized 1 and 5 minutes after birth. The 5 minute score is useful in determining infant morbidity and mortality risk.
  units on a scale | 9 [7 to 9] | 9 [8 to 10] | 9 [7 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Intention to Practice Skin-to-skin Contact After Birth
Description: Both groups will be asked a short survey at the time of admission:
  * their intention to practice skin to skin at the time of delivery
  * if they participated in skin to skin in a previous pregnancy
  * if they had any formal education about skin to skin
  * if they did have formal education was it either
    * a.) Provided at a prenatal appointment
    * b.) A formal class led by either a nurse or a lactation consultant Group B will watch a short video about skin-to-skin contact and will be then reasked a question regarding their intention to practice skin-to-skin contact after birth. This information will allow us to determine if video education impacts the intention to practice skin-to-skin contact after birth.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - no Video Group | Group B - Video Group
Number analyzed (Participants) | 120 | 120
Participants
  Pre-Intervention (video) | 100 | 107
  Post-Intervention | NA — Did not have intervention. | 118

2. Primary Outcome: Actual Practice of Skin-to-skin Contact After Birth
Description: For both video and non-video groups, skin to skin duration (minutes) after delivery will be calculated. The time in minutes from delivery to initiation of skin to skin contact is also collected. This information will allow us to determine if video education impacts the actual practice of skin-to-skin contact after birth.
Time Frame: 1 week
Measure: Median (Full Range); unit: minutes
Arm/Group | Group A - no Video Group | Group B - Video Group
Number analyzed (Participants) | 120 | 120
minutes
  Delivery to Skin to Skin Contact | 6 [0 to 39] | 3 [0 to 26]
  Skin to Skin Duration | 88 [17 to 161] | 91 [13 to 210]

3. Post Hoc Outcome: Number of Participants With Formal Education About Skin to Skin Contact
Description: Measuring formal education training about skin to skin contact prior to admission, provided at either a prenatal appointment or a formal class led by either a nurse or a lactation consultant.
Time Frame: Prior to admission for delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - no Video Group | Group B - Video Group
Number analyzed (Participants) | 120 | 120
Participants | 40 | 38

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Group A - no Video Group | Group B - Video Group
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03200925/Prot_SAP_000.pdf